CLINICAL TRIAL: NCT02399813
Title: Phase 2 Study of ADXS11-001 in Subjects With Persistent/Recurrent, Loco-Regional or Metastatic Squamous Cell Carcinoma of the Anorectal Canal
Brief Title: A Phase 2 Study of Axalimogene Filolisbac (ADXS11-001) in Participants With Carcinoma of the Anorectal Canal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advaxis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADXS001-06; 2015-001053-33 (EudraCT Number)
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Results first posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Anal Cancer; Rectal Cancer
MeSH Terms: conditions — Anus Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Axalimogene filolisbac (Experimental): Participants received intravenous (IV) infusion of axalimogene filolisbac administered over 60 minutes every 3 weeks at a dose of 1 x 10^9 colony forming units (cfu) for up to 2 years or until a discontinuation criterion was met (documented progression, unacceptable adverse events, withdrawn due to investigator's discretion, participant withdraws consent, pregnancy or noncompliance with study procedures or treatments). A treatment cycle was defined as 9 weeks in duration.
  Interventions: Drug: Axalimogene filolisbac

INTERVENTIONS:
Drug: Axalimogene filolisbac
  Other Names: ADXS11-001

SUMMARY:
This is a single arm Phase 2 study. Stage 1 and 2 of the study are monotherapy evaluations of ADXS11-001 in 31 and 24 participants, respectively with persistent/recurrent, loco-regional or metastatic squamous cell carcinoma (SCCA) of the anorectal canal that have received at least 1 regimen for the treatment of advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* Must have cancer of the anal canal OR rectal cancer.
* Must have metastatic disease or persistent/recurrent loco-regional disease
* Prior Therapy: may have received <2 regimens for disease in the metastatic setting. At least one line of therapy.
* Be willing and able to provide written informed consent for the trial.
* Be ≥18 years of age on day of signing informed consent.
* Have measurable disease based on response evaluation criteria in solid tumors (RECIST) 1.1
* Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Demonstrate adequate organ function as defined in protocol.
* Females cannot be pregnant or breastfeeding and must take two methods of birth control

Exclusion Criteria:

* Has not recovered (for example, Grade ≤1 or at baseline) from adverse events (AEs), with the exception of alopecia or Grade ≤2 neuropathy, due to a previously administered agent
* Has a diagnosis of immunodeficiency
* Has known additional malignancy that is progressing or requires active treatment. Treatment of an additional malignancy with chemotherapy, immunotherapy, biologic or hormonal therapy must have occurred 2 years prior. Concurrent use of hormones for non-cancer-related conditions (for example, insulin for diabetes and hormone replacement therapy) is acceptable

  * Note: Local treatment of isolated lesions for palliative intent (for example, by local surgery or radiotherapy), basal cell carcinoma of the skin, or squamous cell carcinoma of the skin, or ductal carcinoma in situ of the breast that has/have been surgically cured is acceptable
* Has known active central nervous system metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided the metastases are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to the first dose of study treatment
* Has concurrent unstable or uncontrolled medical condition (example, active uncontrolled systemic infection, poorly controlled hypertension or history of poor compliance with an anti-hypertensive regimen, unstable angina, congestive heart failure, uncontrolled diabetes) or other chronic disease, which in the opinion of the investigator, could compromise the patient or the study
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents

  * Participants with vitiligo or resolved childhood asthma/atopy would be an exception to this rule.
  * Participants that require intermittent use of inhaled steroids, bronchodilators or local steroid injections may be allowed with sponsor approval.
  * Participants with hypothyroidism stable on hormone replacement or Sjorgen's Syndrome will not be excluded from the study
* Has an active infection requiring systemic therapy. Prior to dosing with study treatment(s), the subject must be at least 5 half-lives from their last dose of antibiotic
* Has any other serious or uncontrolled physical or mental condition/disease that, as judged by the investigator, could place the patient at higher risk derived from his/her participation in the study, could confound results of the study, or would be likely to prevent the patient from complying with the requirements of the study or completing the study.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Participant has implanted medical device(s) that pose a high risk for colonization and/or cannot be easily removed (examples, prosthetic joints, artificial heart valves, pacemakers, orthopedic screw[s], metal plate[s], bone graft[s], or other exogenous implant[s]).

  * Note: More common devices and prosthetics which include arterial and venous stents, dental and breast implants and venous access devices (example, Port-a-Cath or Mediport) are permitted. Participants with any other devices or implants must be approved by Sponsor prior to participation
* Any participant currently requiring or anticipated to require tumor necrosis factor (TNF) blocking agent (example: infliximab) therapy for diagnosis of rheumatologic disease or inflammatory bowel disease (e.g., ankylosing spondylitis, Crohn disease, plaque psoriasis, psoriatic arthritis, rheumatoid arthritis or ulcerative colitis
* Participants who are currently receiving or who have received any phosphoinositide 3-kinase (PI3K) inhibitor within 30 days prior to registration
* Participant has a contraindication (example: sensitivity/allergy) to trimethoprim/sulfamethoxazole and ampicillin
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Has known active hepatitis B or hepatitis C
* Has a known allergy to any component of the study treatment(s) formulations
* Has contraindication to administration of non-steroidal anti-inflammatory drugs (NSAIDs)
* Has undergone a major surgery, including surgery for a new artificial implant and/or medical device which is permitted by the protocol, within 6 weeks prior to the initiation of ADXS11-001 treatment

  * Note: If the participant had a major surgery, all toxicities and/or complications from the intervention must have recovered to at least the baseline or Grade 1 prior to the initiation of ADXS11-001 study therapy. Consult with the Sponsor prior to enrolling participants on the study who recently had a major surgery or have a new artificial implant and/or medical device
* In the opinion of the investigator has rapidly progressing disease, OR has life expectancy of <6 months, OR would be unable to receive at least 1 cycle of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Duarte, California
  - New Haven, Connecticut
  - Indiana University, Indianapolis, Indiana
  - Detroit, Michigan
  - St Louis, Missouri
  - Buffalo, New York
  - Durham, North Carolina
  - Fox Chase, Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas

REFERENCES:
- [Result] Eng C, Fakih M, Amin M, Morris V, Hochster HS, Boland PM, Uronis H. A phase II study of axalimogene filolisbac for patients with previously treated, unresectable, persistent/recurrent loco-regional or metastatic anal cancer. Oncotarget. 2020 Apr 14;11(15):1334-1343. doi: 10.18632/oncotarget.27536. eCollection 2020 Apr 14. PMID 32341753

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Axalimogene Filolisbac
Started | 36
Completed | 0
Not Completed | 36
Not completed — Progressive Disease-Radiographic | 2
Not completed — Death | 20
Not completed — Withdrawal by Subject | 3
Not completed — Initiating a Non-Study Cancer Treatment | 4
Not completed — Lost to Follow-up | 2
Not completed — Other than specified | 5

BASELINE CHARACTERISTICS:
Population: All Treated population: Participants who received at least one dose of axalimogene filolisbac.
Groups:
- Axalimogene Filolisbac: Participants received IV infusion of axalimogene filolisbac administered over 60 minutes every 3 weeks at a dose of 1 x 10^9 cfu for up to 2 years or until a discontinuation criterion was met (documented progression, unacceptable adverse events, withdrawn due to investigator's discretion, participant withdraws consent, pregnancy or noncompliance with study procedures or treatments). A treatment cycle was defined as 9 weeks in duration.
Arm/Group | Axalimogene Filolisbac
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best Overall Response According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: Best response was defined as achievement of complete response (CR) or partial response (PR) per RECIST 1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the first dose until progression or death (maximum duration: 68 weeks)
Population: Participants in the All Treated population were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Axalimogene Filolisbac
Number analyzed (Participants) | 36
percentage of participants | 2.8

2. Primary Outcome: Progression Free Survival
Description: Progression free survival was defined as the time from treatment start until disease progression or death whichever occurred earlier. Participants who have not progressed or who are still alive at the time of evaluation will be censored for the analysis. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. Kaplan-Meier method was used for estimating progression free survival.
Time Frame: From the first dose until progression or death (maximum duration: 68 weeks)
Population: Participants in the All Treated population were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axalimogene Filolisbac
Number analyzed (Participants) | 36
months | 2.0 [1.8 to 2.1]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, was also an adverse event.
Time Frame: From the first dose until end of study (maximum duration: 72 weeks)
Population: Participants in the All Treated population were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Axalimogene Filolisbac
Number analyzed (Participants) | 36
Participants | 36

ADVERSE EVENTS:
Time Frame: From the first dose until end of study (maximum duration: 72 weeks)
Description: All Treated population: Participants who received at least one dose of axalimogene filolisbac.
Arm/Group | Axalimogene Filolisbac
All-Cause Mortality (participants affected / at risk) | 22/36
Serious Adverse Events (participants affected / at risk) | 15/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axalimogene Filolisbac (N=36)
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Enterocutaneous fistula (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Disease progression (General disorders) | 1
Oedema peripheral (General disorders) | 1
Cytokine release syndrome (Immune system disorders) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Blood bilirubin increased (Investigations) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Hallucination (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axalimogene Filolisbac (N=36)
Anaemia (Blood and lymphatic system disorders) | 10
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 2
Vision blurred (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain lower (Gastrointestinal disorders) | 1
Anal haemorrhage (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 2
Enterocutaneous fistula (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 21
Oesophagitis (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 3
Retching (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 1
Chills (General disorders) | 25
Disease progression (General disorders) | 1
Fatigue (General disorders) | 14
Generalised oedema (General disorders) | 1
Hypothermia (General disorders) | 1
Influenza like illness (General disorders) | 2
Non-cardiac chest pain (General disorders) | 4
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 3
Pyrexia (General disorders) | 20
Cholangitis (Hepatobiliary disorders) | 1
Cytokine Release Syndrome (Immune system disorders) | 5
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 4
Arthropod bite (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 8
Rectal injury (Injury, poisoning and procedural complications) | 1
Stoma site extravasation (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 1
Blood creatine increased (Investigations) | 1
Blood creatinine increased (Investigations) | 8
Blood lactate dehydrogenase increased (Investigations) | 1
Body temperature increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Transaminases increased (Investigations) | 2
Weight decreased (Investigations) | 4
White blood cell count decreased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 5
Lactic acidosis (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 9
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 14
Hypersomnia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Abnormal dreams (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Chronic kidney disease (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Swelling face (Skin and subcutaneous tissue disorders) | 1
Embolism (Vascular disorders) | 1
Flushing (Vascular disorders) | 2
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 17
Thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall seek the Sponsor's written approval for study results publication which shall not be unreasonably withheld. Such publication by Institution and/or Investigator may be no earlier than after a cooperative publication has been published with Sponsor or 1 year from date of completion or termination of the Study & only after review and comment by Sponsor. Institution agrees to provide Sponsor a copy of proposed publication at least 60 days prior to submission to a publisher.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT02399813/Prot_SAP_000.pdf